CLINICAL TRIAL: NCT04763317
Title: Precision Medicine in the Prostate Cancer Care Pathway: an Evaluation of Integrating Germline Genetic Testing Into the Management of Men at Risk of / Living With Prostate Cancer
Brief Title: Precision Medicine in the Prostate Cancer Care Pathway
Acronym: PMPRC
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4948
Record Dates: First submitted 2020-09-28; First posted 2021-02-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Genetic Predisposition
MeSH Terms: conditions — Prostatic Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood DNA or Saliva sample is collected from the participant for genetic analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AFFECTED: 1. Affected with PrCa <60 years
  2. Affected with metastatic castration resistant PrCa (mCRPC) or aggressive PrCa (Gleason 4+4 or higher <70 years
  3. Affected with PrCa and a family history defined as three or more cases any age (FDR or SDR)
  Interventions: Genetic: Prostate cancer risk gene panel
- UNAFFECTED (Cohort now closed, recruitment complete): - Aged >30 and with a family history defined as::
  1. FDR diagnosed < 70
  2. 2 or more cases in First or Second Degree Relatives (FDR/SDR) with one case diagnosed < 70 years
  3. 3 or more cases at any age (on same side of family)
  Interventions: Genetic: Prostate cancer risk gene panel

INTERVENTIONS:
Genetic: Prostate cancer risk gene panel — A list of genes created by study experts, thought to increase the risk of prostate cancer from from review previous research, this list is regularly reviewed for accuracy

SUMMARY:
This study aims to evaluate the use of a prostate cancer specific predisposition genetic panel test in men with / at high risk of prostate cancer. The genetic test will analyse men's DNA samples for the presence of mutations in rare genes as well as common genetic variation to provide men with information about their risk of prostate cancer. This study will evaluate the clinical impact of the test on risk assessment and clinical management in terms of screening and treatment.

ELIGIBILITY:
Inclusion Criteria:

Affected cohort:

1. Affected with PrCa < 60 years or
2. Affected with metastatic castration resistant PrCa (mCRPC) at any age or Aggressive PrCa Gleason 4+4 or higher <70 years
3. Affected with family history defined as three or more cases any age (FDR or SDR)

Unaffected cohort: (This cohort is no longer recruiting, it has completed recruitment)

Aged >30 and with a family history defined as:

1. FDR diagnosed < 70
2. 2 or more cases in First or Second Degree Relatives (FDR/SDR) with one case diagnosed < 70 years
3. 3 or more cases at any age (on same side of family)

Exclusion Criteria:

* • WHO performance status 4

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are two pathways for men to be approached about this study; first eligible men will be identified and approached by their clinical team in Urology and Uro-Oncology clinics at the Royal Marsden. Second, men already under the care of the Oncogenetics Research team due to their family history of prostate cancer and who meet the eligibility criteria will be given information about the study as deemed appropriate by the research clinician who has been managing their care (Research Nurse or Clinical Research Fellow).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of genetic variation in affected men | Through study completion, an average of 1 year
  To determine the prevalence of prostate cancer (PrCa) specific genetic variation in men with: (a)young onset PrCa; (b) metastatic PrCa; (c) men with PrCa and a family history of PrCa compared with controls.

SECONDARY OUTCOMES:
Prevalence of genetic variation in unaffected men | Through study completion, an average of 1 year
  To determine the prevalence of prostate cancer specific genetic variation in unaffected men with a strong family history of prostate cancer compared with controls.
Prostate Cancer genetic variation on clinical outcome | Through study completion, an average of 1 year
  To determine how prostate cancer specific genetic variation influences clinical outcome in 'high-risk' vs 'low risk' groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hosital,, Sutton, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No